CLINICAL TRIAL: NCT04302844
Title: A Randomized Controlled Trial of Imago Relationship Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Elizabeth A. Hembree, PhD, Associate Professor of Psychology in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 829071
Record Dates: First submitted 2020-02-14; First posted 2020-03-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Relationship Disorder
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent Evaluators are blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imago Relationship Therapy (IRT) (Active Comparator): Couples will receive 12 to 16 Imago relationship therapy sessions (90 minutes each; one session per week) with an experienced and certified Imago Relationship therapist.
  Interventions: Behavioral: Imago Relationship Therapy
- Waitlist with Bibliotherapy followed by Workshop (Active Comparator): Couples will be asked to wait for 12 weeks before receiving any intervention, and will be given a relationship-focused self-help book to read during that time. After 12 weeks and the 12-week assessment has been completed, couples will receive a Getting the Love You Want workshop.
  Interventions: Behavioral: Waitlist with Bibliotherapy followed by Workshop

INTERVENTIONS:
Behavioral: Imago Relationship Therapy — Imago relationship therapy (IRT) involves learning the Imago dialogue process, which helps couples understand more clearly why they and their partners react as they do. Couples practice communicating in a manner that helps them move from reactivity and blame to understanding and empathy. The dialogue is used to transform conflicts into opportunities for healing and growth, and to connect more deeply and effectively with one another. Specific topics of therapy are determined by the couple's needs and goals. In general, the therapist helps them use the Imago dialogue to promote understanding, heal painful emotions, and make requests of one another to change behaviors. In effort to minimize risk of exposure to the virus that causes COVID-19, since the spring of 2020, therapy sessions will be conducted via telehealth, with a HIPAA-compliant audio/visual platform, and with couples at home or in another private place during the therapy sessions and the therapist in his or her office.
  Other Names: Imago Relationship Therapy (IRT)
  Arms: Imago Relationship Therapy (IRT)
Behavioral: Waitlist with Bibliotherapy followed by Workshop — Participants assigned to this group will be asked to wait for 12 weeks before receiving any intervention, and will be given a relationship-focused self-help book to read, with exercises to practice, during that time. After 12 weeks and the 12-week assessment has been completed, couples will attend an educational workshop that provides the principles and communication skills of Imago Relationship Therapy, typically in a weekend format that is usually about 18-20 hours. The workshops, called "Getting the Love You Want (GTLYW)", are led by certified and experienced Imago workshop presenters, and are attended by a group of couples. The workshop includes presentations, discussions, and practice of communication exercises. Participation in the workshops will also be virtual or via telehealth, as described above.
  Arms: Waitlist with Bibliotherapy followed by Workshop

SUMMARY:
The primary goal of this study, A Randomized Controlled Trial of Imago Relationship Therapy, is to evaluate the efficacy of Imago Relationship Therapy, a form of couples therapy.

DETAILED DESCRIPTION:
Imago relationship therapy (IRT; Hendrix, 2008) is an integrative approach to couples therapy that has been practiced and extensively disseminated for more than 30 years. IRT may be delivered through traditional therapy with a couple, or the Imago principles and skills may be taught to couples through the "Getting the Love You Want" Workshop (GTLYW Workshop), a manualized, 2-day, psychoeducational workshop conducted by certified presenters to groups of couples. The present study is a RCT designed to examine the efficacy of IRT for couples experiencing distress in their committed romantic relationships, and to extend the findings of previous research. Seventy-two (72) couples with relationship distress will be recruited for the study. Couples will be randomly assigned to one of two conditions: Imago therapy alone or bibliotherapy, a control condition, in which couples will be given a self-help book on dyadic communication to read during a 12-week waiting period, followed by a GTLYW workshop.

ELIGIBILITY:
Inclusion Criteria:

1. Straight or LGBTQ couples; both members at least 18 years of age
2. Ability to speak and understand, and read and write, in English language
3. Married/cohabitating for a minimum of 1 year
4. Currently experiencing relationship distress
5. Interest in improving relationship satisfaction/have no immediate plans to terminate the relationship
6. Willingness to participate in study procedures via telehealth and access to the equipment and pricacy required to do so.

Exclusion Criteria:

1. Current alcohol or substance dependence (with active use) in one or both partners
2. Serious suicidal ideation and behavior in one or both partners (i.e., ideation with plan or intent)
3. Current physical violence or partner abuse
4. One or both partners currently involved in a secret affair (i.e., the partner is unaware of this relationship)
5. Current couples-focused psychotherapy treatment that is on-going
6. Couple received IRT or GTLYW workshop within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Relationship Quality Interview (RQI) | 3 to 4 months
  The RQI (Lawrence, Barry, Brock, Bunde, Langer, Ro, et al., 2011) is semi-structured, behaviorally anchored individual interview that takes about 60 minutes to administer. The RQI provides an objective assessment of relationship quality as a dynamic dyadic construct across 5 dimensions: (a) quality of emotional intimacy in the relationship, (b) quality of the couple's sexual relationship, (c) quality of support transactions in the relationship, (d) quality of the couple's ability to share power in the relationship, and (e) quality of conflict/problem-solving interactions in the relationship. The RQI will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Marital Adjustment Test (MAT) | 3 to 4 months
  A 15-item self-report questionnaire that measures relationship satisfaction. The scale focuses on issues such as involvement in joint activities, demonstration of affection, frequency of marital complaints, level of loneliness and well-being, and partner agreement on significant issues. The MAT will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.

SECONDARY OUTCOMES:
Change in Dyadic Adjustment Scale (DAS) | 3 to 4 months
  A 32-item self-report inventory designed to measure satisfaction in intimate dyads. It is a commonly used inventory and has good psychometric properties. The 19 items of the DAS that do not overlap with the MAT will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Davis Interpersonal Reactivity Index (IRI) | 3 to 4 months
  The IRI is a 28-item self-report scale that measures both cognitive and affective components of empathy, and consists of four different 7-item subscales, representing different components of interpersonal sensitivity. The IRI is reliable, well validated and widely used (Davis, 1980). The IRI will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Communication Patterns Questionnaire (CPQ) | 3 to 4 months
  The Communication Patterns Questionnaire assesses a person's perceptions of dyadic communication about relationship problems, and yields scores on three subscales: demand/withdraw, criticize/defend, and positive interaction. The CPQ has demonstrated acceptable reliability and validity. The CPQ will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Couple Satisfaction Inventory -16 | 3 to 4 months
  The CSI-16 is a 16-item self-report that measures current degree of relationship satisfaction. Scores can range from 0 to 81. Higher scores indicate higher levels of relationship satisfaction. The scale has good psychometric properties; see Funk, J.L., & Rogge, R.D. (2007). The CSI-16 will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Quick Inventory of Depressive Symptomatology (QIDS SR-16) (Rush, Trivedi, Ibrahim, Carmody, Arnow, Klein, et al., 2003) | 3 to 4 months
  The QIDS SR-16 is a 16-item self-report measure of depression. It has good internal consistency. The QUIDS SR-16 will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in Generalized Anxiety Disorder - 7 (GAD 7; Spitzer, Kroenke, Williams, 2006). | 3 to 4 months
  The GAD 7 is a 7-item scale developed to diagnose generalized anxiety disorders. It has sensitivity of 89% and specificity of 82% and is commonly used as a brief scale with goo reliability and validity. The GAD 7 will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in PROMIS Item Bank v1.1 Emotional Distress - Anger Short form 5a | 3 to 4 months
  The PROMIS - Anger Short form 5a is a 5-item self-report measure of general anger that is part of the NIH-funded PROMIS® (Patient-Reported Outcomes Measurement Information System), a set of validated person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. The PROMIS - Anger scale will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in PROMIS Item Bank v1.0 Global Satisfaction with Sex | 3 to 4 months
  This PROMIS scale is a 5-item self-report measure of sexual functioning that is part of the NIH-funded PROMIS® (Patient-Reported Outcomes Measurement Information System). The PROMIS Satisfaction with Sex scale will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.
Change in PROMIS Item Bank v1.2 Global Health | 3 to 4 months
  This PROMIS scale is a 10-item self-report measure of general health that is part of the NIH-funded PROMIS® (Patient-Reported Outcomes Measurement Information System). The PROMIS Global Health scale will be used to measure change from: pre-randomization to post-intervention or post-waitlist, and from post-intervention or post-waitlist to 3-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Mood and Anxiety Disorders Treatment & Research Program, Philadelphia, Pennsylvania, United States